CLINICAL TRIAL: NCT05269238
Title: Improvement of the Performance of Lumbar Punctures After Training Students With an Augmented Reality SIMulator
Acronym: APLOSIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8074
Record Dates: First submitted 2022-01-14; First posted 2022-03-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Puncture
Keywords: lumbar puncture; simulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group patient (Other): performing lumbar punctures by students with standard training
  Interventions: Other: performing lumbar punctures by students with standard training
- experimental group patient (Experimental): performing lumbar punctures by students with standard training and an augmented reality simulator
  Interventions: Other: training students augmented reality simulator

INTERVENTIONS:
Other: performing lumbar punctures by students with standard training — performance of the puncture by the student have been previously trained with standard training
  Arms: control group patient
Other: training students augmented reality simulator — performance of the puncture by the student have been previously trained using the augmented reality simulator
  Arms: experimental group patient

SUMMARY:
Lumbar punctures (LP) are frequent invasive procedures that are anxiety-provoking for both the patient and the clinicans performing the procedure. LP is performed by many practitioners, whether they are emergency physicians, neurologists, neurosurgeons, internists or rheumatologists. Learning how to perform LP is essentially done at the patient's bed by showing the students how a procedure is performed and then having them perform it directly on a patient afterwards. The recent development of simulation in health care with the credo "never the first time on the patient" requires the development of training devices faithful to reality.

The rheumatology department of the Strasbourg University Hospital has been working for 3 years, in collaboration with the Strasbourg start-up InSimo, on the development of an LP simulator. This simulator is original because it allows the feeling by pressure of the passage of the various structures, and in particular the yellow ligament. This sensation is made possible by a haptic force feedback device.

ELIGIBILITY:
Inclusion criteria:

* Requiring a lumbar puncture as part of their routine care
* Male or female of legal age with no upper age limit
* French speaking
* Subject affiliated to a social health insurance scheme
* Not having expressed his or her opposition to the re-use of his or her data in the context of this research

Exclusion criteria:

* Previously undergone a lumbar puncture
* BMI > 35 kg/m².
* Spinal ankylosis: history of ankylosing spondylitis or Forestier's disease
* Impossible to give the subject informed information (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Subject under court protection
* Subject under guardianship or curatorship
* Contraindication to the use of Emlapatch

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Success rate of lumbar punctures in patients according to whether the students performing their first lumbar puncture were previously trained to perform this invasive procedure using the augmented reality simulator versus standard teaching. | 3 days
  Success rate of lumbar puncture as assessed by the collection of cerebrospinal fluid (CSF) at the end of the procedure. A successful LP is defined as the collection of CSF at the end of the procedure performed by the student without the assistance of a senior physician or resident and without interruption of the procedure by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Felten R, Bigaut K, Wirth T, Kremer L, Gauer L, Arnold C, Ollivier I, Godet J, Scherlinger M, Dubois M, Sebbag E, De Seze J, Gottenberg JE. Advancing medical training with augmented reality and haptic feedback simulator: outcomes of a randomized controlled trial on lumbar puncture. BMC Med Educ. 2025 Aug 30;25(1):1231. doi: 10.1186/s12909-025-07536-6. PMID 40885925